CLINICAL TRIAL: NCT02031471
Title: TOSCARA: An Open-label, Single Arm Study to Evaluate the Efficacy, Safety and Tolerability of Tocilizumab (TCZ) Subcutaneous in TCZ-naïve Patients With Active Rheumatoid Arthritis
Brief Title: TOSCARA Study: A Study of Subcutaneous Tocilizumab (RoActemra/Actemra) in Participants With Active Rheumatoid Arthritis Naïve to RoActemra/Actemra Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28701
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Adults with rheumatoid arthritis received a fixed dose of tocilizumab during the 24-week open-label core study and those entering the long term extension (LTE) period further received a fixed dose up to a maximum of 28 weeks or until tocilizumab was commercially available and/or reimbursed whichever came first. A fixed dose of 162 mg tocilizumab was administered subcutaneously once weekly.
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: tocilizumab — Fixed dose of 162 mg subcutaneously weekly
  Other Names: RoActemra/Actemra

SUMMARY:
This open-label, single-arm study will evaluate the efficacy, safety and tolerability of subcutaneously administered tocilizumab in monotherapy and/or in combination with methotrexate and other non-biologic disease modifying anti-rheumatic drug (DMARDs) in participants with active rheumatoid arthritis (RA) who are naïve to tocilizumab. Participants will receive tocilizumab 162 milligram (mg) subcutaneously weekly for 24 weeks. Participants who complete the core study achieving at least a moderate European League Against Rheumatism (EULAR) response at Week 24 may enter the extension phase and receive for a further 28 weeks at the most.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Active moderate to severe rheumatoid arthritis according to the revised (1987) American College of Rheumatology (ACR) criteria or EULAR/ACR (2010) criteria
* Inadequate response or intolerant to previous therapy with two or more non-biologic disease-modifying anti-rheumatic drugs (DMARDs), one of which is methotrexate, administered in an optimal way during at least 3 months; eligible participants may also be inadequate responders to a maximum of one biologic DMARD
* Oral corticosteroids (</= 10 milligram per day (mg/day) prednisolone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs; up to the recommended dose) are permitted if on stable dose regimen for >/= 4 weeks prior to baseline
* Permitted DMARDs are allowed if at stable dose for at least 4 weeks prior to baseline
* Receiving treatment on an outpatient basis, not including tocilizumab
* Females of childbearing potential and males with female partners of childbearing potential must agree to use reliable means of contraception as defined by protocol

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline or during long term extension (LTE) period
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16
* Prior history of or current inflammatory joint disease other than RA
* Exposure to tocilizumab (intravenous or subcutaneous) at any time prior to baseline
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Intraarticular or parenteral corticosteroids within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Evidence of serious concomitant disease or disorder
* Known active current or history of recurrent infection
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active Tuberculosis (TB) requiring treatment within the previous 3 years
* Positive for hepatitis B or hepatitis C
* Primary or secondary immunodeficiency (history of or currently active)
* Pregnant or lactating women
* Neuropathies or other conditions that might interfere with pain evaluation
* Inadequate hematologic, renal or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Belgium (14):
  - Aalst
  - Assebroek
  - Bonheiden
  - Brussels
  - Genk
  - Ghent
  - Gilly (Charleroi)
  - Gosselies
  - Haine-Saint-Paul
  - Liège
  - Roeselare
  - Sijsele
  - Sint-Niklaas
  - Wilrijk
- Luxembourg, Luxembourg

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 62 participants were screened, 57 participants were enrolled. Participants who completed the 24 Week Treatment Period achieving at least a moderate European League Against Rheumatism (EULAR) response at Week 24 were allowed to enter the Long Term Extension (LTE) Period.
Groups:
- Tocilizumab: Adults with rheumatoid arthritis received a fixed dose of tocilizumab during the 24-week open-label core study and those entering the long term extension (LTE) period further received a fixed dose up to a maximum of 28 weeks or until tocilizumab was commercially available and/or reimbursed whichever came first. Participants entered 8 weeks of follow-up either at the end of the 24-week open-label core study or after completion of the LTE. A fixed dose of 162 milligram (mg) tocilizumab was administered subcutaneously once weekly.
Period: 24 Week Treatment Period
Arm/Group | Tocilizumab
Started | 57
Completed | 46
Not Completed | 11
Not completed — Adverse Event | 6
Not completed — Participant Decision to Withdraw | 2
Not completed — Protocol Violation | 1
Not completed — Insufficient Therapeutic Response | 1
Not completed — Hypersensitivity Reaction | 1
Period: Long Term Extension (LTE) Period
Arm/Group | Tocilizumab
Started | 39 (Only participants who achieved at least a moderate EULAR response at Week 24 entered the LTE Period.)
Completed | 37
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Insufficient Therapeutic Response | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab.
Groups:
- Tocilizumab: Adults with rheumatoid arthritis received a fixed dose of tocilizumab during the 24-week open-label core study and those entering the LTE period further received a fixed dose up to a maximum of 28 weeks or until tocilizumab was commercially available and/or reimbursed whichever came first. A fixed dose of 162 mg tocilizumab was administered subcutaneously once weekly.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.49 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28 - Erythrocyte Sedimentation Rate (DAS28-ESR) Score in the Full Analysis Set (FAS)
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count of 28 joints (TJC28), swollen joint count of 28 joints (SJC28), patient's global assessment of disease activity visual analog scale (PGA VAS) with 0=no disease activity to 100=maximum disease activity displayed on the 100-millimeter (mm) horizontal VAS and acute phase reactant (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]) for a total possible score of 0 to 10. For this study ESR was used to calculate the DAS28 score. The index is calculated using the following formula: DAS28 = (0.56*√[TJC28]) + (0.28*√[SJC28]) + (0.70*ln[ESR]) + (0.014*VAS). Higher scores represent higher disease activity. A negative change from baseline indicates an improvement.
Time Frame: From baseline to Week 24
Population: The FAS consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab. Here n is the number of participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=56) | 5.55 (1.17)
  Change at Week 24 (n=42) | -3.24 (1.47)

2. Primary Outcome: Change From Baseline in Disease Activity Score 28 - Erythrocyte Sedimentation Rate (DAS28-ESR) Score in the Per Protocol Set (PPS)
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC28, SJC28, PGA VAS with 0=no disease activity to 100=maximum disease activity displayed on the 100-mm horizontal VAS and acute phase reactant (ESR or CRP) for a total possible score of 0 to 10. For this study ESR was used to calculate the DAS28 score. The index is calculated using the following formula: DAS28 = (0.56*√[TJC28]) + (0.28*√[SJC28]) + (0.70*ln[ESR]) + (0.014*VAS). Higher scores represent higher disease activity. A negative change from baseline indicates an improvement.
Time Frame: From baseline to Week 24
Population: The PPS consisted of all participants of the FAS having a value at baseline and at Week 24 for the endpoint DAS28-ESR, excluding sponsor defined deviation(s) which could have affected the evaluation of the primary endpoint (DAS28-ESR). Here, n is the number of participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n= 27) | 5.73 (1.33)
  Change at Week 24 (n= 20) | -3.21 (1.42)

3. Secondary Outcome: Percentage of Participants With Positive American College of Rheumatology (ACR) Response Scores
Description: The ACR core set of outcome measures and their definition of improvement includes a >= 20% improvement (ACR20) compared to Baseline in both SJC and TJC as well as in three out of five additional parameters: Physician's Global Assessment of disease activity VAS, PGA VAS, patient's assessment of pain VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI), and acute phase reactant (CRP or ESR). VAS range for all assessments was 0=no disease activity to 100=maximum disease activity displayed on the 100-mm horizontal VAS. Achievement of an ACR50 requires a >= 50% improvement in the same parameters and an ACR70 requires a >= 70% improvement.
Time Frame: From Baseline to Week 2, Week 24, and Week 52
Population: The FAS consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab. Here, n is the number of participants with evaluable data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Baseline: ACR 20 (n=55) | 0
  Week 2: ACR 20 (n=51) | 21.6
  Week 24: ACR 20 (n=39) | 84.6
  Week 52: ACR 20 (n=8) | 100
  Baseline: ACR 50 (n=55) | 0
  Week 2: ACR 50 (n=52) | 1.9
  Week 24: ACR 50 (n=39) | 66.7
  Week 52: ACR 50 (n=8) | 62.5
  Baseline: ACR 70 (n=55) | 0
  Week 2: ACR 70 (n=52) | 0
  Week 24: ACR 70 (n=39) | 38.5
  Week 52: ACR 70 (n=8) | 25.0

4. Secondary Outcome: Percentage of Participants With Responses According to European League Against Rheumatism (EULAR ) Criteria
Description: EULAR response was calculated as the difference between DAS28-ESR scores at baseline and Week 24, and reported as the percentage of participants with good, moderate, or no response. Good responders = decrease from baseline >1.2 with a DAS28 score of <=3.2; moderate responders = decrease from baseline >1.2 with a DAS28 score of >3.2, or decrease from baseline >0.6 to <=1.2 with a DAS28 score of <=5.1; non-responders = decrease from baseline <=0.6 or decrease from baseline >0.6 and <=1.2 with a DAS28 score of >5.1.
Time Frame: From Baseline to Week 2, Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Week 2: Good response (n=56) | 17.9
  Week 24: Good response (n=42) | 76.2
  Week 2: Moderate response (n=56) | 50.0
  Week 24: Moderate response (n=42) | 19.0
  Week 2: No response (n=56) | 32.1
  Week 24: No response (n=42) | 4.8

5. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)/Clinical Disease Activity Index (CDAI)
Description: SDAI is a similar index to DAS28 but has the advantage of not needing a complicated mathematical formula for its determination, but a simple arithmetical addition of TJC28 and SJC28, PGA VAS and Physician Global Assessment of disease activity VAS, and CRP concentration in mg/L. CDAI does not incorporate an acute response, therefore it can be used to evaluate disease activity in the absence of laboratory testing of CRP and ESR. VAS range for all assessments was 0=no disease activity to 100=maximum disease activity displayed on the 100-mm horizontal VAS. SDAI scores ranged from 0 to 86, CDAI from 0 to 76 with higher scores indicating increased disease activity. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=53) | 33.26 (13.50)
  Change at Week 2: SDAI (n=52) | -9.00 (11.89)
  Change at Week 24: SDAI (n=38) | -25.33 (13.63)
  Change at Week 52: SDAI (n=7) | -34.04 (16.01)
  Baseline: CDAI (n= 55) | 31.86 (12.60)
  Change at Week 2: CDAI (n=55) | -7.61 (11.51)
  Change at Week 24: CDAI (n=42) | -23.55 (13.03)
  Change at Week 52: CDAI (n=8) | -29.99 (13.89)

6. Secondary Outcome: Change in Total Tender/Swollen Joint Counts (TJC/SJC)
Description: An assessment of 66 joints for swelling and 68 joints for tenderness was made. Joints were assessed and classified as swollen/not swollen and tender/not tender by pressure and joint manipulation on physical examination. Joint prosthesis, arthrodesis or fused joints were not taken into consideration for swelling or tenderness. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Joint Counts
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Joint Counts
  Baseline: TJC (n=53) | 16.02 (11.77)
  Change at Week 2: TJC (n=53) | -3.58 (8.91)
  Change at Week 24: TJC (n=41) | -12.10 (11.07)
  Change at Week 52: TJC (n=8) | -17.25 (13.02)
  Baseline: SJC (n=55) | 10.20 (7.14)
  Change at Week 2: SJC (n=55) | -3.93 (7.33)
  Change at Week 24: SJC (n=42) | -9.81 (7.84)
  Change at Week 52: SJC (n=8) | -11.75 (7.76)

7. Secondary Outcome: Percentage of Participants With Corticosteroid Dose Reduction/Discontinuation
Time Frame: Up to Week 52
Population: The FAS consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 26
percentage of participants | 50.0

8. Secondary Outcome: Percentage of Participants Achieving CDAI Remission, CDAI Low Disease Activity, Moderate Disease Activity and High Disease Activity
Description: CDAI is calculated by simple arithmetical addition of TJC28 and SJC28, PGA VAS and Physician Global Assessment of disease activity VAS. VAS range was 0=no disease activity to 100=maximum disease activity displayed on the 100-mm horizontal VAS. Total CDAI score ranges from 0 to 76 with higher scores indicating increased disease activity. Clinical remission = score ≤ 2.8; Low disease activity = score > 2.8 and ≤ 10.0; Moderate disease activity = score > 10.0 and ≤ 22.0; High disease activity = score > 22.0.
Time Frame: Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Baseline: Clinical remission (n=55) | 0
  Week 2: Clinical remission (n=56) | 1.8
  Week 24: Clinical remission (n=43) | 30.2
  Week 52: Clinical remission (n=8) | 37.5
  Baseline: Low disease activity (n=55) | 0
  Week 2: Low disease activity (n=56) | 7.1
  Week 24: Low disease activity (n=43) | 34.9
  Week 52: Low disease activity (n=8) | 25.0
  Baseline: Moderate disease activity (n=55) | 21.8
  Week 2: Moderate disease activity (n=56) | 48.2
  Week 24: Moderate disease activity (n=43) | 30.2
  Week 52: Moderate disease activity (n=8) | 37.5
  Baseline: High disease activity (n=55) | 78.2
  Week 2: High disease activity (n=56) | 42.9
  Week 24: High disease activity (n=43) | 4.7
  Week 52: High disease activity (n=8) | 0

9. Secondary Outcome: Percentage of Participants Achieving SDAI Remission, SDAI LDA, Moderate Disease Activity and High Disease Activity
Description: SDAI is calculated by simple arithmetical addition of TJC28 and SJC28, PGA VAS and Physician Global Assessment of disease activity VAS, and CRP concentration in mg/L. VAS range was 0=no disease activity to 100=maximum disease activity displayed on the 100-mm horizontal VAS. Total SDAI score ranges from 0 to 86 with higher scores indicating increased disease activity. Clinical remission = score ≤ 3.3; Low disease activity = score > 3.3 and ≤ 11.0; Moderate disease activity = score > 11.0 and ≤ 26.0; high disease activity = score > 26.0.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Baseline: Clinical remission (n=53) | 0
  Week 2: Clinical remission (n=55) | 1.8
  Week 24: Clinical remission (n=40) | 30.0
  Week 52: Clinical remission (n=7) | 42.9
  Baseline: Low disease activity (n=53) | 0
  Week 2: Low disease activity (n=55) | 7.3
  Week 24: Low disease activity (n=40) | 40.0
  Week 52: Low disease activity (n=7) | 14.3
  Baseline: Moderate disease activity (n=53) | 30.2
  Week 2: Moderate disease activity (n=55) | 54.5
  Week 24: Moderate disease activity (n=40) | 25.0
  Week 52: Moderate disease activity (n=7) | 42.9
  Baseline: High disease activity (n=53) | 69.8
  Week 2: High disease activity (n=55) | 36.4
  Week 24: High disease activity (n=40) | 5.0
  Week 52: High disease activity (n=7) | 0

10. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Remission, DAS28-ESR LDA, Moderate Disease Activity and High Disease Activity
Description: The DAS28 score is a measure of the participant's disease activity calculated using TJC28, SJC28, PGA VAS with 0=no disease activity to 100=maximum disease activity displayed on the 100-millimeter (mm) horizontal VAS and acute phase reactant (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]) for a total possible score of 0 to 10. For this study ESR was used to calculate the DAS28 score. The index is calculated using the following formula: DAS28 = (0.56*√[TJC28]) + (0.28*√[SJC28]) + (0.70*ln[ESR]) + (0.014*VAS). Higher scores represent higher disease activity. Clinical remission = score <2.6; Low disease activity = score ≥2.6 and ≤3.2; Moderate disease activity = score > 3.2 and ≤5.1; High disease activity = score >5.1.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Baseline: Clinical remission (n=56) | 0
  Week 2: Clinical remission (n=56) | 7.1
  Week 24: Clinical remission (n=42) | 64.3
  Week 52: Clinical remission (n=8) | 87.5
  Baseline: Low disease activity (n=56) | 1.8
  Week 2: Low disease activity (n=56) | 16.1
  Week 24: Low disease activity (n=42) | 16.7
  Week 52: Low disease activity (n=8) | 0
  Baseline: Moderate disease activity (n=56) | 35.7
  Week 2: Moderate disease activity (n=56) | 53.6
  Week 24: Moderate disease activity (n=42) | 19.0
  Week 52: Moderate disease activity (n=8) | 12.5
  Baseline: High disease activity (n=56) | 62.5
  Week 2: High disease activity (n=56) | 23.2
  Week 24: High disease activity (n=42) | 0
  Week 52: High disease activity (n=8) | 0

11. Secondary Outcome: Percentage of Participants Achieving a Clinically Significant Improvement in DAS28
Description: The DAS28 score is a measure of the participant's disease activity calculated using TJC28, SJC28, PGA VAS with 0=no disease activity to 100=maximum disease activity displayed on the 100-millimeter (mm) horizontal VAS and acute phase reactant (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]) for a total possible score of 0 to 10. For this study ESR was used to calculate the DAS28 score. The index is calculated using the following formula: DAS28 = (0.56*√[TJC28]) + (0.28*√[SJC28]) + (0.70*ln[ESR]) + (0.014*VAS). Higher scores represent higher disease activity. DAS28 Clinically Significant Improvement was defined as a DAS28 score reduction of at least 1.2 units from Baseline.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Week 2 (n=56) | 66.1
  Week 24 (n=42) | 90.5
  Week 52 (n=8) | 100

12. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity VAS
Description: Physician's Global Assessment of disease activity VAS represents the physician's assessment of the participant's current disease activity on a 100 mm horizontal VAS. The extreme left end of the line represents 0= "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end 100= "maximum disease activity". This was completed by the Treating Physician (or designee). A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=56) | 64.93 (17.73)
  Change at Week 2 (n=56) | -16.34 (16.88)
  Change at Week 24 (n=45) | -48.93 (25.06)
  Change at Week 52 (n=9) | -57.44 (23.26)

13. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity VAS
Description: PGA VAS represents the participant's overall assessment of their current disease activity on a 100 mm horizontal VAS. The extreme left end of the line represents 0= "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end 100="maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 67.28 (22.25)
  Change at Week 2 (n=57) | -11.82 (23.23)
  Change at Week 24 (n=46) | -36.02 (29.38)
  Change at Week 52 (n=9) | -44.78 (35.87)

14. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain VAS
Description: Patient's Assessment of Pain VAS represents the participant's assessment of his/her current level of pain on a 100 mm horizontal VAS. The extreme left end of the line represents 0="no pain" and the extreme right end 100="unbearable pain". A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 66.77 (21.43)
  Change at Week 2 (n=57) | -11.32 (19.74)
  Change at Week 24 (n=46) | -35.37 (27.03)
  Change at Week 52 (n=9) | -49.33 (39.58)

15. Secondary Outcome: Acute Phase Reactants: Change From Baseline in CRP
Description: A negative change from baseline in CRP level indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
milligrams per liter (mg/L)
  Baseline (n=55) | 13.79 (20.78)
  Change at Week 2 (n=54) | -13.19 (20.64)
  Change at Week 24 (n=42) | -10.12 (14.50)
  Change at Week 52 (n=8) | -25.07 (23.03)

16. Secondary Outcome: Acute Phase Reactants: Change From Baseline in ESR
Description: A negative change from baseline in ESR indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters per hour (mm/hr)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
millimeters per hour (mm/hr)
  Baseline (n=56) | 33.75 (28.90)
  Change at Week 2 (n=55) | -19.95 (18.22)
  Change at Week 24 (n=44) | -22.80 (24.88)
  Change at Week 52 (n=9) | -27.78 (23.82)

17. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The Stanford HAQ-DI is a patient-oriented outcome assessment questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities. Each category contains multiple questions, which were answered using a 4-point scale from 0 to 3. The overall index score was an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 1.44 (0.68)
  Change at Week 2 (n=57) | -0.08 (0.43)
  Change at Week 24 (n=46) | -0.54 (0.68)
  Change at Week 52 (n=9) | -1.33 (0.68)

18. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: The symptom-specific measure FACIT-F was developed to assess chronic illness therapy with special emphasis on fatigue in the past 7 days. In this study, only the FACIT-F short questionnaire, which is a shorter version of the initial FACIT-F questionnaire, was used. Each of the questions is categorically answered using the scales 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. The figures are reversed during score calculations, so that higher score values indicate more favorable conditions. The 13 items included in the FACIT-F short can be used to calculate the brief score for FACIT-F scale (score range: 0-52). A positive change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 26.09 (10.75)
  Change at Week 2 (n=57) | 2.32 (9.58)
  Change at Week 24 (n=45) | 10.53 (12.06)
  Change at Week 52 (n=9) | 20.89 (12.35)

19. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The participant self-rates each of these seven areas of sleep. Scoring of answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. Global scores range from 0 to 21 and a global sum of "5" or greater indicates a "poor" sleeper. Although there are several questions that request the evaluation of the participant's bed mate or roommate, these are not scored. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 4, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 8.81 (4.39)
  Change at Week 4 (n=54) | -1.24 (3.53)
  Change at Week 24 (n=46) | -2.63 (4.14)
  Change at Week 52 (n=9) | -4.56 (5.88)

20. Secondary Outcome: Change From Baseline in Patient Quality of Sleep VAS
Description: The Patient Quality of Sleep VAS assessment represents the participant's assessment of his/her current quality of sleep on a 100 mm horizontal VAS. The extreme left end of the line represents 0="no difficulty to sleep" and the extreme right end 100="extreme sleeping difficulties". A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 54.95 (31.23)
  Change at Week 2 (n=57) | -8.40 (23.72)
  Change at Week 24 (n=46) | -21.93 (30.87)
  Change at Week 52 (n=9) | -34.22 (37.03)

21. Secondary Outcome: Change From Baseline in Arthritis Impact Measurement Scale-Short Form (AIMS-SF)
Description: The AIMS-SF is a reduced version of the validated AIMS2 questionnaire. The Short Form has been developed using a comprehensive expert-based approach and supported by psychometric testing. The AIMS-SF is a self-administered questionnaire to measure changes in global health, pain, mobility and social function in adult patients with arthritis and reports scores for physical, symptoms, affect, social and work assessments. Scores range from 0 to 10, higher scores indicating higher impact of arthritis on the assessments. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 4, Week 24 and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline: Physical (n= 49) | 3.57 (1.92)
  Change at Week 4: Physical (n= 47) | -0.57 (1.36)
  Change at Week 24: Physical (n=38) | -1.41 (1.83)
  Change at Week 52: Physical (n=3) | -3.62 (2.23)
  Baseline: Symptom (50) | 6.33 (2.59)
  Change at Week 4: Symptom (n= 48) | -1.15 (2.46)
  Change at Week 24: Symptom (n=40) | -2.69 (2.80)
  Change at Week 52: Symptom (n=3) | -3.89 (5.91)
  Baseline: Affect (n=50) | 5.07 (2.22)
  Change at Week 4: Affect (n= 48) | -0.66 (1.56)
  Change at Week 24: Affect (n=40) | -1.74 (2.22)
  Change at Week 52: Affect (n=3) | -4.50 (2.22)
  Baseline: Social (n=50) | 5.36 (1.73)
  Change at Week 4: Social (n= 48) | 0.18 (1.41)
  Change at Week 24: Social (n=40) | -0.56 (1.61)
  Change at Week 52: Social (n=3) | -1.46 (2.37)
  Baseline: Work (n=26) | 3.17 (2.46)
  Change at Week 4: Work (n= 23) | -0.92 (2.53)
  Change at Week 24: Work (n=21) | -0.65 (2.87)
  Change at Week 52: Work (n=1) | 3.75 (NA) — Standard deviation is not estimable for 1 participant.

22. Secondary Outcome: Change From Baseline in Patient Fatigue VAS
Description: The Patient Fatigue VAS assessment represents the participant's assessment of his/her current level of fatigue on a 100 mm horizontal VAS. The extreme left end of the line represents 0="no fatigue" and the extreme right end 100="extreme fatigue". A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=57) | 60.19 (24.79)
  Change at Week 2 (n=57) | -3.74 (20.68)
  Change at Week 24 (n=46) | -21.48 (28.07)
  Change at Week 52 (n=9) | -50.89 (26.11)

23. Secondary Outcome: Change From Baseline in Patient Satisfaction VAS
Description: The Patient Satisfaction VAS assessment represents the participant's assessment of his/her current satisfaction with treatment on a 100 mm horizontal VAS. The extreme left end of the line represents 0="no satisfaction" and the extreme right end 100="extremely satisfied". A positive change from baseline indicates an improvement.
Time Frame: From Baseline to Week 2, Week 24 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=53) | 39.66 (28.63)
  Change at Week 2 (n=53) | 9.49 (33.97)
  Change at Week 24 (n=43) | 33.07 (35.50)
  Change at Week 52 (n=8) | 49.38 (35.12)

24. Secondary Outcome: Change From Baseline in Work Instability Scale for Rheumatoid Arthritis (RA-WIS)
Description: The 23-item RA-WIS is a simple, validated screening tool for work instability, i.e., the consequences of a mismatch between an individual's functional ability and their work tasks. This self-administered questionnaire covers a broad range of specific work-related issues and enables monitoring the risk of work disability in rheumatoid arthritis patients. The RA-WIS is scored by summing responses from all 23 scale items. The scale ranges from 0 to 23. Cut points have been established to differentiate levels of work instability: low < 10, moderate 10-17 and high > 17. A negative change from baseline indicates an improvement.
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Baseline (n=26) | 13.15 (6.05)
  Change at Week 24 (n=22) | -3.55 (6.96)

25. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM ) Scores
Description: The abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) derived from the TSQM Version 1.4 but without the five items of the side effects domain, is a reliable and valid measure to assess participants' satisfaction with treatment. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain. Domains included are effectiveness, convenience and global satisfaction.
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
Units on a scale
  Effectiveness (n=46) | 66.7 (19.07)
  Convenience (n=46) | 76.09 (15.66)
  Global Satisfaction (n=46) | 65.06 (15.52)

26. Secondary Outcome: Safety: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 52 weeks
Population: The FAS consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants | 96.5

27. Secondary Outcome: Safety: Percentage of Participants With Anti-tocilizumab Antibodies
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  Baseline (n= 55) | 0
  Week 24 (n= 43) | 1.7

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: The safety population consisted of all participants included in the study who received at least one dose of subcutaneous tocilizumab.
Groups:
- Tocilizumab: Adults with rheumatoid arthritis received a fixed dose of tocilizumab during the 24-week open-label core study and those entering the long term extension (LTE) period further received a fixed dose up to a maximum of 28 weeks or until tocilizumab was commercially available and/or reimbursed whichever came first. A fixed dose of 162 milligram (mg) tocilizumab was administered subcutaneously once weekly.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 5/57
Other Adverse Events (participants affected / at risk) | 36/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=57)
Atrial Flutter (Cardiac disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Arthritis Infective (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=57)
Vertigo (Ear and labyrinth disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Injection site erythema (General disorders) | 3
Bronchitis (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.